CLINICAL TRIAL: NCT00000723
Title: Chemotherapy, Radiotherapy, and Azidothymidine for AIDS-Related Primary CNS Lymphoma
Brief Title: The Use of Chemotherapy Plus Radiotherapy Plus Azidothymidine in Patients With AIDS-Related Lymph Node Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 009; 10985 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Lymphoma; Methotrexate; Leucovorin; Dexamethasone; Drug Evaluation; Drug Therapy, Combination; Combined Modality Therapy; Acquired Immunodeficiency Syndrome; Zidovudine; Brain Neoplasms
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; AIDS-Related Opportunistic Infections; Lymphoma; Acquired Immunodeficiency Syndrome; Brain Neoplasms | interventions — Methotrexate; Leucovorin; Zidovudine; Dexamethasone

INTERVENTIONS:
Drug: Methotrexate
Drug: Leucovorin calcium
Drug: Zidovudine
Drug: Dexamethasone

SUMMARY:
To determine the safety and toxicity of high-dose systemic methotrexate (MTX) and dexamethasone (DEX) combined with zidovudine (AZT) and brain irradiation in patients with AIDS-related primary central nervous system (CNS) lymphoma and to determine response rates and survival of treated patients. Also to determine if the treatment inhibits HIV replication in patients who are HIV culture and/or antigen positive and to assess the incidence of opportunistic infection in these patients Results of radiation given to patients with AIDS-related high-grade CNS lymphoma have been disappointing, with short survival times due to infection complications. However, complete response has been documented after radiation in some patients. High-dose MTX will be used to improve the possibility of a greater antineoplastic response than that obtained by radiation alone. Since the underlying immunodeficiency state is not affected by therapy directed against the lymphoma, patients are still prone to life-threatening opportunistic infections or relapse of lymphomatous disease within the CNS. Accordingly, AZT will also be used in an attempt to alter the overall natural history of the disease.

DETAILED DESCRIPTION:
Results of radiation given to patients with AIDS-related high-grade CNS lymphoma have been disappointing, with short survival times due to infection complications. However, complete response has been documented after radiation in some patients. High-dose MTX will be used to improve the possibility of a greater antineoplastic response than that obtained by radiation alone. Since the underlying immunodeficiency state is not affected by therapy directed against the lymphoma, patients are still prone to life-threatening opportunistic infections or relapse of lymphomatous disease within the CNS. Accordingly, AZT will also be used in an attempt to alter the overall natural history of the disease.

Radiation begins on day 1 of therapy. Patients receive dexamethasone orally (PO) or by intravenous injection (IV) on days 1-10. MTX IV over 6 hours weekly for a total of 4 doses starts 1 week after completion of the cranial radiation. Leucovorin (LCV) IV or PO begins 6 hours after MTX has been completed over 6 hours for 8 doses. AZT while awake starts on day 1 of therapy and continues for 52 weeks. Patients are reevaluated with computerized tomography (CT) or magnetic resonance imaging (MRI) scan of the brain at conclusion of radiation therapy and systemic treatment, 6 and 10 weeks respectively. If there is a complete or partial response (CR or PR), patient will remain on study and continue to receive AZT; if stable disease or no response, patient will be taken off study. Reevaluation at 16 weeks from start of study will be done. If CR or PR, the patient will continue AZT for 1 year. If there is no change or progression of disease, or if the patient develops evidence of systemic lymphomatous disease, patient will be taken off study.

ELIGIBILITY:
Inclusion Criteria

* Patient must have negative titers for toxoplasmosis or other infectious etiology for CNS disease.

Prior Medication:

Allowed:

* Zidovudine may be continued per protocol specifications.

Exclusion Criteria

* Pathologic diagnosis of lymphoma in central nervous system (CNS) must be confirmed but no previous treatment is allowed. In participating institutions where CNS biopsies cannot be obtained, the patient may be considered eligible if space-occupying lesions have been demonstrated on computerized tomography or magnetic resonance imaging with negative titers for toxoplasmosis or negative response to empiric therapy for intracerebral toxoplasmosis and negative workup for other infectious etiology of CNS disease.

Co-existing Condition:

Patients with the following are excluded:

* Positive titers for toxoplasmosis. Positive titers for other infectious etiology of CNS disease. Acute intercurrent infection. A second active tumor other than nonmelanomatous skin cancer or Kaposi's sarcoma. Lymphomatous meningitis alone without a mass lesion in the brain.

Concurrent Medication:

Excluded:

* Acetaminophen, nonsteroidal anti- inflammatory agents, and corticosteroids other than dexamethasone.

Prior Medication:

Excluded:

* Acetaminophen, nonsteroidal anti-inflammatory agents, and corticosteroids other than dexamethasone.
* Excluded within 2 weeks of study entry:
* Immunomodulating agents.
* Excluded within 30 days of study entry:
* Any investigational agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Study Completion 1990-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levine AM, Study Chair
Locations (1):
- Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana, United States